CLINICAL TRIAL: NCT02304302
Title: Phase II Multicenter 16-Week Randomized Double Blind Placebo-Controlled Evaluation of the Efficacy, Tolerability and Safety of Memantine Hydrochloride on Enhancing the Cognitive Abilities of Adolescents and Young Adults With Down Syndrome
Brief Title: Down Syndrome Memantine Follow-up Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Alana USA Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 121971
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-04

CONDITIONS: Down Syndrome; Intellectual Disability
Keywords: Memantine; Episodic Memory; CVLT; Hippocampus dependent memory; Short-term memory
MeSH Terms: conditions — Down Syndrome; Intellectual Disability | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Identically-looking placebo pills to memantine will be dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Interventions: Drug: Placebo
- Memantine (Experimental): Memantine will be dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Encapsulated Namenda 10 mg bid (after four-week standard dose titration protocol)
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — Identically looking placebo capsules bid (after a four-week regimen designed to mimic standard dose titration protocol)
  Other Names: Inactive Capsules
  Arms: Placebo

SUMMARY:
The purpose of this research study is to learn if the medication Memantine Hydrochloride (the study medication) can help adolescents and young adults with Down syndrome. Dr. Alberto Costa and his research team want to see if a 16-week treatment with this medication can improve the participant's ability to learn and remember things. In this study, memantine hydrochloride will be used. Thus, the researchers want to learn whether the study drug can help improve memory in young adults with Down syndrome. To test the effect of the study medicine, half of the people in the study will receive the study medicine and half will receive a placebo (an inactive substance). Memantine is an approved medication to treat memory and thinking problems in persons with Alzheimer disease. However, little is known about the effect of this medication in persons with Down syndrome and it has not been approved for use in persons with Down syndrome.

DETAILED DESCRIPTION:
This study seeks to investigate if the medication Memantine Hydrochloride can help young adults with Down syndrome. Two hundred persons with Down syndrome from both genders and between 15 and 32 years of age will be recruited from two sites: Cleveland, OH, USA and São Paulo, SP, Brazil. Participants will be assigned randomly to either a placebo group or a group taking the active medication with a 50% probability of being on either group. Neither the participants nor the investigators will know who will be taking the study medication and who will be taking the placebo during the study. Only the investigational pharmacist will have access to this information.

Up to 60 people with Down syndrome of the recruited study participants will take part on an optional magnetic resonance imaging (MRI) study. This investigation is aimed at helping to make the EEG study more precise and to find out whether the study medication has any significant effect on the structure of the brain.

Additionally, we will recruit a control group of 60 age- and gender-matched participants without Down syndrome. The goal is to investigate how different groups of people activate their brains when they hear or see something, and if he can use high-density EEG and MRI to see how this study medication works in persons with Down syndrome. In other words, this additional control group should help us ascertain which parts of the test results are due to a person having Down syndrome and which ones are not. Persons without Down syndrome will only come for one EEG visit and one MRI visit, and not be asked to take the study medication.

The visits for the participants with Down syndrome will be as follows:

Screening visit (approximately 2-hour long). The subject will be asked about his/her health, medical history, social background, and work background, as well as some simple questions to determine performance on tests of memory and function that are part of this study. Informed consent and assent will be obtained in this visit. At the end of this visit, an EEG machine will be used to access brain responses to different auditory and visual stimuli. Some will be asked if they would be willing to have an MRI performed, but this portion is not imperative.

A urine sample will be collected and used to obtain cells that will be kept frozen for potential future studies. If the date of the screening visit is not convenient, this sample can be collected during any of the next five visits.

Visit 1 (approximately 1 hour). Pulse, blood pressure, and an electrocardiogram (ECG) will be taken. At the end of the visit, urine and blood samples will be taken. Pregnancy will also be checked.

Visit 2 (2-3 hours). Tests of memory, learning, and reasoning skills will be conducted before the start of the study medicine or placebo. At the end of this visit, a 60-day supply of either the study medicine or the placebo will be given. This will need to be taken for 16 weeks.

Visit 3 (approximately 30 minutes). Eight weeks after the beginning of the treatment, the participant will return to assess how she/he is doing under the treatment. Pulse, blood pressure, a physical exam, and pregnancy will be checked. At this visit, another supply of study medicine will be given.

Visit 4 (2-3 hours). Sixteen weeks after starting the medicine, the participant will take a second series of tests in learning, memory, and reasoning skills to find out whether there were any changes in these skills.

Visit 5 (approximately 1 hour). In the 16th or 17th week after starting the medicine, the participant will meet one more time with the doctor from visits 1 and 3. Vital signs, a physical exam, and an ECG will be taken, as well as a blood sample to ensure nothing has changed with the participant's general health. For women, a pregnancy test will be performed.

If for some reason the subject withdraws from this study prior to Visit 5, he/she will be asked to return to the clinic for a "Treatment Discontinuation Visit." In addition, if the participant discontinues the medication prior to the end of the study, he/she will be asked to complete a "Retrieved Dropout Visit" on the date that should have represented Visit 5. Study medication will not be provided beyond the study period.

ELIGIBILITY:
Inclusion Criteria:

* Cytogenetically documented Trisomy 21 or Complete Unbalanced Translocation of Chromosome 21. Mosaic Trisomy 21 and partial translocations will be excluded from the study
* No pregnancy by serum testing at screening. Females of child-bearing potential, sexually active must be practicing a reliable method of birth control. Urine pregnancy tests will be done at the 2 follow-up medical visits
* Laboratory findings within normal limits or judged clinically insignificant at baseline
* Vital signs within normal limits for age. Stable, medically treated hypotension will be allowed
* ECG must demonstrate predominately normal sinus rhythm. Minor abnormalities documented as clinically insignificant will be allowed
* Participants and their authorized representatives will provide written informed consent
* Participants who have received any experimental drug for Down syndrome must undergo a washout
* All participants must: Be in general good health as judged by the investigators; Be able to swallow oral medication; Have a reliable caregiver or family member who agrees to accompany participant to all visits, provide information about the participant as required by the protocol, and ensure compliance with the medication schedule; Be sufficiently proficient in English (USA) or Portuguese (Brazil) to reliably complete the study assessments
* Age and gender matching participants without Down syndrome, must be: Males or females without Down syndrome aged-matching (within 3 years) participants with Down syndrome whom they are expected to serve as controls

Exclusion Criteria:

* Participant weighing less than 40 kg
* Current psychiatric or neurologic diagnosis other than Down syndrome (e.g., major depressive disorder, schizophrenia, bipolar disorder, autism, Alzheimer disease)
* Current treatment with psychotropic drugs
* Drug or alcohol abuse or dependence
* Significant suicide risk or who would require treatment with electro-convulsive therapy or with psychotropic drugs during the study or who have received treatment with a depot neuroleptic drug within 6 months of entering the study.
* Current or expected (within the next 6 months) hospitalization or residence in a skilled nursing facility (may reside in group homes or other residential settings with no skilled nursing)
* Active or clinically significant conditions affecting absorption, distribution, or metabolism of study drug (e.g. inflammatory bowel disease or celiac disease)
* Significant allergies to or other significant intolerance of memantine therapy, its ingredients, or with contraindications to memantine therapy as stated in the prescribing information
* Participants who are expected to require general anesthetics during the course of the study
* Presence or recent history of seizure disorder (< 3 years).
* Clinically significant and/or clinically unstable systemic disease. (Those with controlled hypothyroidism must be on a stable dose of medication for at least 3 months prior to screening and have normal serum T-4 and TSH at screening; and those with controlled diabetes mellitus must have an HbA1c of < 8.0% and a random serum glucose value of < 170 mg/dl)
* Severe infections or a major surgical operation within 3 months prior to screening
* History of persistent cognitive deficits immediately following head trauma.
* Donation of blood or blood products less that 30 days prior to screening, while participating in the study, or four weeks after completion of the study
* Inability to comply with the protocol or perform the outcomes measures due to significant hearing or visual impairment or other issues judged relevant by the investigators
* Exclusion criteria for controls without Down syndrome: History of substance abuse, major psychiatric disorder, attention deficit disorder, or learning disability; Beck Depression Score greater than 10; Exclusion criteria specific to MR scanning; Pregnancy; Neurologic history

Ages: 15 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2014-10; Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto C Costa, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center; Stephen L Ruedrich, MD, Study Director — University Hospitals Cleveland Medical Center
Locations (2):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States
- Sociedade Beneficente Israelita Brasileira Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Abbeduto L, Pavetto M, Kesin E, Weissman MD, Karadottir S, O'Brien A, Cawthon S. The linguistic and cognitive profile of Down syndrome: evidence from a comparison with fragile X syndrome. Downs Syndr Res Pract. 2001 Oct;7(1):9-15. doi: 10.3104/reports.109. PMID 11706811
- [Background] Bittles AH, Glasson EJ. Clinical, social, and ethical implications of changing life expectancy in Down syndrome. Dev Med Child Neurol. 2004 Apr;46(4):282-6. doi: 10.1017/s0012162204000441. No abstract available. PMID 15077706
- [Background] Boada R, Hutaff-Lee C, Schrader A, Weitzenkamp D, Benke TA, Goldson EJ, Costa AC. Antagonism of NMDA receptors as a potential treatment for Down syndrome: a pilot randomized controlled trial. Transl Psychiatry. 2012 Jul 17;2(7):e141. doi: 10.1038/tp.2012.66. PMID 22806212
- [Background] Brock J, Jarrold C. Serial order reconstruction in Down syndrome: evidence for a selective deficit in verbal short-term memory. J Child Psychol Psychiatry. 2005 Mar;46(3):304-16. doi: 10.1111/j.1469-7610.2004.00352.x. PMID 15755306
- [Background] Carr J. Six weeks to twenty-one years old: a longitudinal study of children with Down's syndrome and their families. Third Jack Tizard memorial lecture. J Child Psychol Psychiatry. 1988 Jul;29(4):407-31. doi: 10.1111/j.1469-7610.1988.tb00734.x. PMID 2975288
- [Background] Carr J. Stability and change in cognitive ability over the life span: a comparison of populations with and without Down's syndrome. J Intellect Disabil Res. 2005 Dec;49(Pt 12):915-28. doi: 10.1111/j.1365-2788.2005.00735.x. PMID 16287480
- [Background] Chen KH, Reese EA, Kim HW, Rapoport SI, Rao JS. Disturbed neurotransmitter transporter expression in Alzheimer's disease brain. J Alzheimers Dis. 2011;26(4):755-766. doi: 10.3233/JAD-2011-110002. PMID 21743130 (Retraction: PMID 27814301 J Alzheimers Dis. 2016 Nov 1;55(1):445)
- [Background] Chez MG, Burton Q, Dowling T, Chang M, Khanna P, Kramer C. Memantine as adjunctive therapy in children diagnosed with autistic spectrum disorders: an observation of initial clinical response and maintenance tolerability. J Child Neurol. 2007 May;22(5):574-9. doi: 10.1177/0883073807302611. PMID 17690064
- [Background] Costa AC, Scott-McKean JJ. Prospects for improving brain function in individuals with Down syndrome. CNS Drugs. 2013 Sep;27(9):679-702. doi: 10.1007/s40263-013-0089-3. PMID 23821040
- [Background] Costa AC, Scott-McKean JJ, Stasko MR. Acute injections of the NMDA receptor antagonist memantine rescue performance deficits of the Ts65Dn mouse model of Down syndrome on a fear conditioning test. Neuropsychopharmacology. 2008 Jun;33(7):1624-32. doi: 10.1038/sj.npp.1301535. Epub 2007 Aug 15. PMID 17700645
- [Background] Danysz W, Parsons CG. Alzheimer's disease, beta-amyloid, glutamate, NMDA receptors and memantine--searching for the connections. Br J Pharmacol. 2012 Sep;167(2):324-52. doi: 10.1111/j.1476-5381.2012.02057.x. PMID 22646481
- [Background] Erickson CA, Mullett JE, McDougle CJ. Open-label memantine in fragile X syndrome. J Autism Dev Disord. 2009 Dec;39(12):1629-35. doi: 10.1007/s10803-009-0807-3. Epub 2009 Jul 16. PMID 19609663
- [Background] Erickson CA, Posey DJ, Stigler KA, Mullett J, Katschke AR, McDougle CJ. A retrospective study of memantine in children and adolescents with pervasive developmental disorders. Psychopharmacology (Berl). 2007 Mar;191(1):141-7. doi: 10.1007/s00213-006-0518-9. Epub 2006 Oct 3. PMID 17016714
- [Background] Fernandez G, Weyerts H, Schrader-Bolsche M, Tendolkar I, Smid HG, Tempelmann C, Hinrichs H, Scheich H, Elger CE, Mangun GR, Heinze HJ. Successful verbal encoding into episodic memory engages the posterior hippocampus: a parametrically analyzed functional magnetic resonance imaging study. J Neurosci. 1998 Mar 1;18(5):1841-7. doi: 10.1523/JNEUROSCI.18-05-01841.1998. PMID 9465008
- [Background] Findling RL, McNamara NK, Stansbrey RJ, Maxhimer R, Periclou A, Mann A, Graham SM. A pilot evaluation of the safety, tolerability, pharmacokinetics, and effectiveness of memantine in pediatric patients with attention-deficit/hyperactivity disorder combined type. J Child Adolesc Psychopharmacol. 2007 Feb;17(1):19-33. doi: 10.1089/cap.2006.0044. PMID 17343551
- [Background] Francis PT, Palmer AM, Snape M, Wilcock GK. The cholinergic hypothesis of Alzheimer's disease: a review of progress. J Neurol Neurosurg Psychiatry. 1999 Feb;66(2):137-47. doi: 10.1136/jnnp.66.2.137. PMID 10071091
- [Background] Hanney M, Prasher V, Williams N, Jones EL, Aarsland D, Corbett A, Lawrence D, Yu LM, Tyrer S, Francis PT, Johnson T, Bullock R, Ballard C; MEADOWS trial researchers. Memantine for dementia in adults older than 40 years with Down's syndrome (MEADOWS): a randomised, double-blind, placebo-controlled trial. Lancet. 2012 Feb 11;379(9815):528-36. doi: 10.1016/S0140-6736(11)61676-0. Epub 2012 Jan 10. PMID 22236802
- [Background] Hosenbocus S, Chahal R. Memantine: a review of possible uses in child and adolescent psychiatry. J Can Acad Child Adolesc Psychiatry. 2013 May;22(2):166-71. PMID 23667364
- [Background] Hu NW, Ondrejcak T, Rowan MJ. Glutamate receptors in preclinical research on Alzheimer's disease: update on recent advances. Pharmacol Biochem Behav. 2012 Feb;100(4):855-62. doi: 10.1016/j.pbb.2011.04.013. Epub 2011 Apr 22. PMID 21536064
- [Background] Jarrold C, Baddeley AD, Hewes AK. Verbal short-term memory deficits in Down syndrome: a consequence of problems in rehearsal? J Child Psychol Psychiatry. 2000 Feb;41(2):233-44. PMID 10750549
- [Background] Javitt DC, Steinschneider M, Schroeder CE, Arezzo JC. Role of cortical N-methyl-D-aspartate receptors in auditory sensory memory and mismatch negativity generation: implications for schizophrenia. Proc Natl Acad Sci U S A. 1996 Oct 15;93(21):11962-7. doi: 10.1073/pnas.93.21.11962. PMID 8876245
- [Background] Kaindl AM, Degos V, Peineau S, Gouadon E, Chhor V, Loron G, Le Charpentier T, Josserand J, Ali C, Vivien D, Collingridge GL, Lombet A, Issa L, Rene F, Loeffler JP, Kavelaars A, Verney C, Mantz J, Gressens P. Activation of microglial N-methyl-D-aspartate receptors triggers inflammation and neuronal cell death in the developing and mature brain. Ann Neurol. 2012 Oct;72(4):536-49. doi: 10.1002/ana.23626. PMID 23109148
- [Background] Kew JN, Kemp JA. Ionotropic and metabotropic glutamate receptor structure and pharmacology. Psychopharmacology (Berl). 2005 Apr;179(1):4-29. doi: 10.1007/s00213-005-2200-z. Epub 2005 Feb 25. PMID 15731895
- [Background] Kornhuber J, Kennepohl EM, Bleich S, Wiltfang J, Kraus T, Reulbach U, Meineke I. Memantine pharmacotherapy: a naturalistic study using a population pharmacokinetic approach. Clin Pharmacokinet. 2007;46(7):599-612. doi: 10.2165/00003088-200746070-00005. PMID 17596105
- [Background] Korostenskaja M, Nikulin VV, Kicic D, Nikulina AV, Kahkonen S. Effects of NMDA receptor antagonist memantine on mismatch negativity. Brain Res Bull. 2007 May 30;72(4-6):275-83. doi: 10.1016/j.brainresbull.2007.01.007. Epub 2007 Feb 2. PMID 17452287
- [Background] Leverenz JB, Raskind MA. Early amyloid deposition in the medial temporal lobe of young Down syndrome patients: a regional quantitative analysis. Exp Neurol. 1998 Apr;150(2):296-304. doi: 10.1006/exnr.1997.6777. PMID 9527899
- [Background] Li S, Mallory M, Alford M, Tanaka S, Masliah E. Glutamate transporter alterations in Alzheimer disease are possibly associated with abnormal APP expression. J Neuropathol Exp Neurol. 1997 Aug;56(8):901-11. doi: 10.1097/00005072-199708000-00008. PMID 9258260
- [Background] Li S, Hong S, Shepardson NE, Walsh DM, Shankar GM, Selkoe D. Soluble oligomers of amyloid Beta protein facilitate hippocampal long-term depression by disrupting neuronal glutamate uptake. Neuron. 2009 Jun 25;62(6):788-801. doi: 10.1016/j.neuron.2009.05.012. PMID 19555648
- [Background] Lieberman DN, Mody I. Regulation of NMDA channel function by endogenous Ca(2+)-dependent phosphatase. Nature. 1994 May 19;369(6477):235-9. doi: 10.1038/369235a0. PMID 7514273
- [Background] Lockrow J, Boger H, Bimonte-Nelson H, Granholm AC. Effects of long-term memantine on memory and neuropathology in Ts65Dn mice, a model for Down syndrome. Behav Brain Res. 2011 Aug 10;221(2):610-22. doi: 10.1016/j.bbr.2010.03.036. Epub 2010 Apr 2. PMID 20363261
- [Background] Marczynski TJ. GABAergic deafferentation hypothesis of brain aging and Alzheimer's disease; pharmacologic profile of the benzodiazepine antagonist, flumazenil. Rev Neurosci. 1995 Jul-Sep;6(3):221-58. doi: 10.1515/revneuro.1995.6.3.221. PMID 8717636
- [Background] Naatanen R. The mismatch negativity: a powerful tool for cognitive neuroscience. Ear Hear. 1995 Feb;16(1):6-18. PMID 7774770
- [Background] Naatanen R. Mismatch negativity (MMN) as an index of central auditory system plasticity. Int J Audiol. 2008 Nov;47 Suppl 2:S16-20. doi: 10.1080/14992020802340116. PMID 19012108
- [Background] Parker SE, Mai CT, Canfield MA, Rickard R, Wang Y, Meyer RE, Anderson P, Mason CA, Collins JS, Kirby RS, Correa A; National Birth Defects Prevention Network. Updated National Birth Prevalence estimates for selected birth defects in the United States, 2004-2006. Birth Defects Res A Clin Mol Teratol. 2010 Dec;88(12):1008-16. doi: 10.1002/bdra.20735. Epub 2010 Sep 28. PMID 20878909
- [Background] Parsons CG, Stoffler A, Danysz W. Memantine: a NMDA receptor antagonist that improves memory by restoration of homeostasis in the glutamatergic system--too little activation is bad, too much is even worse. Neuropharmacology. 2007 Nov;53(6):699-723. doi: 10.1016/j.neuropharm.2007.07.013. Epub 2007 Aug 10. PMID 17904591
- [Background] Patterson D, Costa AC. Down syndrome and genetics - a case of linked histories. Nat Rev Genet. 2005 Feb;6(2):137-47. doi: 10.1038/nrg1525. No abstract available. PMID 15640809
- [Background] Pennington BF, Moon J, Edgin J, Stedron J, Nadel L. The neuropsychology of Down syndrome: evidence for hippocampal dysfunction. Child Dev. 2003 Jan-Feb;74(1):75-93. doi: 10.1111/1467-8624.00522. PMID 12625437
- [Background] Petrides M, Milner B. Deficits on subject-ordered tasks after frontal- and temporal-lobe lesions in man. Neuropsychologia. 1982;20(3):249-62. doi: 10.1016/0028-3932(82)90100-2. PMID 7121793
- [Background] Picton TW, Alain C, Otten L, Ritter W, Achim A. Mismatch negativity: different water in the same river. Audiol Neurootol. 2000 May-Aug;5(3-4):111-39. doi: 10.1159/000013875. PMID 10859408
- [Background] Roizen NJ, Patterson D. Down's syndrome. Lancet. 2003 Apr 12;361(9365):1281-9. doi: 10.1016/S0140-6736(03)12987-X. PMID 12699967
- [Background] Rueda N, Llorens-Martin M, Florez J, Valdizan E, Banerjee P, Trejo JL, Martinez-Cue C. Memantine normalizes several phenotypic features in the Ts65Dn mouse model of Down syndrome. J Alzheimers Dis. 2010;21(1):277-90. doi: 10.3233/JAD-2010-100240. PMID 20421694
- [Background] Sani G, Serra G, Kotzalidis GD, Romano S, Tamorri SM, Manfredi G, Caloro M, Telesforo CL, Caltagirone SS, Panaccione I, Simonetti A, Demontis F, Serra G, Girardi P. The role of memantine in the treatment of psychiatric disorders other than the dementias: a review of current preclinical and clinical evidence. CNS Drugs. 2012 Aug 1;26(8):663-90. doi: 10.2165/11634390-000000000-00000. PMID 22784018
- [Background] Scott-McKean JJ, Costa AC. Exaggerated NMDA mediated LTD in a mouse model of Down syndrome and pharmacological rescuing by memantine. Learn Mem. 2011 Nov 18;18(12):774-8. doi: 10.1101/lm.024182.111. Print 2011 Dec. PMID 22101180
- [Background] Seow D, Gauthier S. Pharmacotherapy of Alzheimer disease. Can J Psychiatry. 2007 Oct;52(10):620-9. doi: 10.1177/070674370705201003. PMID 18020110
- [Background] Seung HK, Chapman R. Digit span in individuals with Down syndrome and in typically developing children: temporal aspects. J Speech Lang Hear Res. 2000 Jun;43(3):609-20. doi: 10.1044/jslhr.4303.609. PMID 10877432
- [Background] Swainson R, Hodges JR, Galton CJ, Semple J, Michael A, Dunn BD, Iddon JL, Robbins TW, Sahakian BJ. Early detection and differential diagnosis of Alzheimer's disease and depression with neuropsychological tasks. Dement Geriatr Cogn Disord. 2001 Jul-Aug;12(4):265-80. doi: 10.1159/000051269. PMID 11351138
- [Background] Tayeb HO, Yang HD, Price BH, Tarazi FI. Pharmacotherapies for Alzheimer's disease: beyond cholinesterase inhibitors. Pharmacol Ther. 2012 Apr;134(1):8-25. doi: 10.1016/j.pharmthera.2011.12.002. Epub 2011 Dec 16. PMID 22198801
- [Background] Tikhonravov D, Neuvonen T, Pertovaara A, Savioja K, Ruusuvirta T, Naatanen R, Carlson S. Dose-related effects of memantine on a mismatch negativity-like response in anesthetized rats. Neuroscience. 2010 Jun 2;167(4):1175-82. doi: 10.1016/j.neuroscience.2010.03.014. Epub 2010 Mar 15. PMID 20298759
- [Background] Tilleux S, Hermans E. Neuroinflammation and regulation of glial glutamate uptake in neurological disorders. J Neurosci Res. 2007 Aug 1;85(10):2059-70. doi: 10.1002/jnr.21325. PMID 17497670
- [Background] Turner S, Alborz A. Academic attainments of children with Down's syndrome: a longitudinal study. Br J Educ Psychol. 2003 Dec;73(Pt 4):563-83. doi: 10.1348/000709903322591244. PMID 14713378
- [Background] Turner S, Alborz A, Gayle V. Predictors of academic attainments of young people with Down's syndrome. J Intellect Disabil Res. 2008 May;52(Pt 5):380-92. doi: 10.1111/j.1365-2788.2007.01038.x. Epub 2008 Jan 14. PMID 18205756
- [Background] Umbricht D, Schmid L, Koller R, Vollenweider FX, Hell D, Javitt DC. Ketamine-induced deficits in auditory and visual context-dependent processing in healthy volunteers: implications for models of cognitive deficits in schizophrenia. Arch Gen Psychiatry. 2000 Dec;57(12):1139-47. doi: 10.1001/archpsyc.57.12.1139. PMID 11115327
- [Background] Vicari S, Marotta L, Carlesimo GA. Verbal short-term memory in Down's syndrome: an articulatory loop deficit? J Intellect Disabil Res. 2004 Feb;48(Pt 2):80-92. doi: 10.1111/j.1365-2788.2004.00478.x. PMID 14723651
- [Background] Vicari S, Caselli MC, Gagliardi C, Tonucci F, Volterra V. Language acquisition in special populations: a comparison between Down and Williams syndromes. Neuropsychologia. 2002;40(13):2461-70. doi: 10.1016/s0028-3932(02)00083-0. PMID 12417473
- [Background] Zigman W, Schupf N, Haveman M, Silverman W. The epidemiology of Alzheimer disease in intellectual disability: results and recommendations from an international conference. J Intellect Disabil Res. 1997 Feb;41 ( Pt 1):76-80. doi: 10.1111/j.1365-2788.1997.tb00679.x. PMID 9089462
- [Background] Zigman WB, Lott IT. Alzheimer's disease in Down syndrome: neurobiology and risk. Ment Retard Dev Disabil Res Rev. 2007;13(3):237-46. doi: 10.1002/mrdd.20163. PMID 17910085
- [Background] Costa AC. Alzheimer disease: Treatment of Alzheimer disease in Down syndrome. Nat Rev Neurol. 2012 Mar 13;8(4):182-4. doi: 10.1038/nrneurol.2012.40. No abstract available. PMID 22410580
- [Background] Choi DW. Excitotoxic cell death. J Neurobiol. 1992 Nov;23(9):1261-76. doi: 10.1002/neu.480230915. PMID 1361523
- [Background] Brandão IM, V. F, R. MR (2012) Prevalence of People with Down Syndrome in Brazil. In: Scientia Plena (www.scientiaplena.org.br).
- [Background] Pueschel SM, Hopmann MR (1993) Speech and language abilities of children with Down syndrome. In: Enhancing children's communication: Research foundations for intervention (Kaisen AP, Gray DB, eds), pp 335-362. London: Brookes.
- [Result] Costa ACS, Brandao AC, Boada R, Barrionuevo VL, Taylor HG, Roth E, Stasko MR, Johnson MW, Assir FF, Roberto MP, Salmona P, Abreu-Silveira G, Bederman I, Prendergast E, Huls A, Abrishamcar S, Mustacchi Z, Scheidemantel T, Roizen NJ, Ruedrich S. Safety, efficacy, and tolerability of memantine for cognitive and adaptive outcome measures in adolescents and young adults with Down syndrome: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2022 Jan;21(1):31-41. doi: 10.1016/S1474-4422(21)00369-0. PMID 34942135

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Identically-looking placebo capsules to memantine were dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Placebo: Identically looking placebo capsules bid (after a four-week regimen designed to mimic standard dose titration protocol)
- Memantine: Memantine capsules were dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Memantine: Encapsulated Memantine 10 mg bid (after four-week standard dose titration protocol)
Period: Overall Study
Arm/Group | Placebo | Memantine
Started | 79 | 81
Completed | 76 | 73
Not Completed | 3 | 8
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 4
Not completed — Removed from analysis due to low medication compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Identically looking placebo capsules to memantine were dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Placebo: Identically looking placebo capsules bid (after a four-week regimen designed to mimic standard dose titration protocol)
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (4.2) | 20.4 (4.7) | 20.35 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 36 | 38 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67
  Brazil | 47 | 46 | 93
Mother's Years of Education [Mean (Standard Deviation); unit: Years of education] | 14.6 (3.9) | 14.4 (3.8) | 14.5 (3.8)
Father's Years of Education [Mean (Standard Deviation); unit: Years of education] | 13.8 (4.3) | 14.5 (3.9) | 14.3 (4.1)
Hypothyroidism [Count of Participants; unit: Participants] | 37 | 41 | 78
Obesity [Count of Participants; unit: Participants] | 24 | 25 | 49
Sleep apnea [Count of Participants; unit: Participants] | 11 | 13 | 24
Diabetes [Count of Participants; unit: Participants] | 0 | 3 | 3
California Verbal Learning Test Second Edition-Short Form (CVLT-II-sf) total free recall score [Mean (Standard Deviation); unit: units on a scale] — The primary efficacy measure is focused on episodic memory. The CVLT-II short form assesses supraspan word learning ability as an index of episodic verbal long-term memory. We hypothesize that treatment with memantine will produce significant improvements in this test. The main dependent variable selected, based on prior literature was the total number of target items correct summed across learning trials 1-4. Scale Range: from 0 to 36; higher scores represent higher cognitive functioning.
  units on a scale | 14.2 (7.1) | 12.8 (6.4) | 13.5 (6.7)
Matrices Subtest of the Differential Ability Scales-II (DAS-II) [Mean (Standard Deviation); unit: units on a scale] — This test provides a measure of non-verbal reasoning ability that requires subjects to visually inspect a matrix of 4 or 9 pictures that has a missing piece. Participants infer a rule or pattern in the stimuli and select the appropriate response from a range of 4-6 possibilities. Since age norms are not available for individuals older than 17y11m, the ability score was used. This score based on Rasch modeling that corrects for different items sets being administered to participants. The minimum value of the DAS-II Score is 0 and the maximum is 153. Higher values represent a better outcome.
  units on a scale | 51.5 (12.3) | 51.4 (13.4) | 51.4 (12.9)
Scales of Independent Behavior-Revised (SIB-R) broad independence standard score [Mean (Standard Deviation); unit: units on a scale] — This is a measure of adaptive functioning that integrates information from 13 different domains (e.g., gross motor, social interaction, eating, toileting, dressing, personal self-care, etc.). It is in a questionnaire format, which a caregiver can complete while the participant is being tested. The minimum value of the SIB-R Score Scale in this study was -24 (this number is below 0 because -24 was the minimum value for the worst performing participant in the trial) and the maximum value of this scale is 153; higher scores mean higher adaptive functioning.
  units on a scale | 45.9 (25.7) | 43 (22.8) | 44.4 (23.2)
Peabody Picture Vocabulary Test-IV (PPVT-IV) [Mean (Standard Deviation); unit: units on a scale] — This is a measure of receptive semantics. The participant is asked to point to a picture (out of 4) that corresponds to a word spoken by the examiner. As this test has a 0.85 correlation with composite measures of Verbal IQ (i.e. from the Wechsler Intelligence Scale series), it can be used to estimate overall intellectual functioning. The total number of items correct was used as the dependent variable, following the administration manual's rules for basals and ceilings. The minimum value for this scale is 0 and the maximum value is 192, higher scores mean higher intellectual functioning.
  units on a scale | 46.6 (20.7) | 45.4 (18.6) | 46 (19.7)
Level of intellectual disability (Severe) [Count of Participants; unit: Participants] | 22 | 30 | 52
Level of intellectual disability (Moderate) [Count of Participants; unit: Participants] | 29 | 25 | 54
Level of intellectual disability (Mild to typical) [Count of Participants; unit: Participants] | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the California Verbal Learning Test-II (CVLT-II) Short Form Total Free Recall
Description: The primary efficacy measure is focused on episodic memory. The CVLT-II short form assesses supraspan word learning ability as an index of episodic verbal long-term memory. We hypothesize that treatment with memantine will produce significant improvements in this test. The main dependent variable selected, based on prior literature was the total number of target items correct summed across learning trials 1-4. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2). Scale Range: from 0 to 36; higher scores represent better outcomes.
Time Frame: baseline and 16 weeks from start of treatment
Population: The analysis population consisted of participants who completed 16 weeks of treatment and had neuropsychological assessments at baseline (T1) and after treatment (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Identically looking placebo pills to memantine were dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Placebo: Identically looking placebo capsules bid (after a four-week regimen designed to mimic standard dose titration protocol)
- Memantine: Memantine were dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Memantine: Encapsulated Memantine 10 mg bid (after four-week standard dose titration protocol)
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 3.3 (5.15) | 3.49 (4.5)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.61, Mixed Models Analysis; Mean Difference (Net) = 0.34, 95% CI 2-sided [-0.98 to 1.67]

2. Secondary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the Paired Associates Learning (PAL) From the Cambridge Neuropsychological Test Automated Battery (CANTAB)
Description: This is a measure of non-verbal memory that requires the participant to learn associations between an abstract visual pattern and its location. Two dependent variables have been selected: Total number of items correct on the first trial of each stage, and total number of stages completed. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2). The minimum value of the PAL Memory Score Scale is 0 and the maximum value is 21; higher scores mean better outcomes.
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 1 (3.76) | 0.67 (3.83)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.57, Mixed Models Analysis; Mean Difference (Net) = -0.32, 95% CI 2-sided [-1.43 to 0.80]

3. Secondary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the Recall of Digits Forward (From the Differential Ability Scales; DAS-II)
Description: This is a measure of rote short-term verbal memory. Total number of items correct were used as the dependent variable. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2). The minimum value for this scale is 0 and the maximum value is 38; higher scores mean a better outcome.
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 0.03 (2.37) | -0.01 (1.93)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.91, Mixed Models Analysis; Median Difference (Net) = -0.04, 95% CI 2-sided [-0.74 to 0.66]

4. Secondary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the Pattern Recognition Memory (PRM; Part of the Cambridge Neuropsychological Test Automated Battery -- CANTAB)
Description: This is a measure of non-verbal memory. Total number correct across the two series of items presented was used as the dependent variable. We used the PRM total scale in this study, which represents the sum of the PRM correct scores (ranging from 0 to 24) and the PRM delayed scores (ranging from 0 to 24). Therefore, the range of the PRM total scale is from 0 to 48; higher values mean better outcomes.
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 0.45 (4.24) | -0.05 (4.48)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.48, Mixed Models Analysis; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-1.91 to 0.91]

5. Secondary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the Spatial Working Memory (Part of the Cambridge Neuropsychological Test Automated Battery -- CANTAB)
Description: The test requires participants to search under a series of colored boxes to locate a "blue token" hidden underneath one of them. During a series of trials, the participant is told that the token will be in a new location each time and that they should not go back to a location he or she has looked in previously. The main dependent variable was the total number of errors ("between errors"), which indexes the number of times a participant went back to a box where a token had already been found, lower scores mean better performance. The minimum value of the Spatial Working Memory scale is 0 and the maximum value is 137 (which was computed as the equivalent to -4 standard deviations from the mean of this measure); higher scores mean worse outcomes. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2).
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | -0.09 (11.99) | -1.4 (11.66)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.50, Mixed Models Analysis; Mean Difference (Net) = -1.31, 95% CI 2-sided [-5.14 to 2.53]

6. Secondary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the Spatial Span (Part of the Cambridge Neuropsychological Test Automated Battery -- CANTAB)
Description: This measure is a computerized version of the Corsi Blocks task, a long-standing neuropsychological test. The main dependent variables selected for this test was the span length, which is the longest sequence of numbers recalled accurately. The minimum value of the Spatial Span Length Score Scale is 0 and the maximum value is 9; higher scores mean better outcomes. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2).
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 0.13 (1.30) | 0.03 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.52 to 0.32]

7. Secondary Outcome: Efficacy of the Drug Memantine as Assessed by Change in Score on the The Go - No Go Task
Description: This is a measure of inhibitory control, often used as a marker for prefrontal-striatal function integrity. Specifically, it measures the participant's ability to inhibit pre-potent behavioral responses that have been established by provision of prior "go" or "no-go" cues in a classical conditioning paradigm. The main dependent variables selected was speed of response of execution to Go targets. The minimum value of the speed of response of execution to Go targets is 280 milliseconds (ms) and the maximum value is 1000 ms; higher scores mean worse outcomes. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2).
Time Frame: baseline and 16 weeks from start of treatment
Population: The analysis population consisted of participants who completed 16 weeks of treatment and had neuropsychological assessments at baseline (T1) and after treatment (T2). Notice that, for this specific test, some participants stopped midway.
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Placebo: Identically-looking placebo pills to memantine will be dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Placebo: Identically looking placebo capsules bid (after a four-week regimen after a four-week regimen designed to mimic standard dose titration protocol)
- Memantine: Memantine will be dispensed in a 66-day supply (56 days plus 10 extra days) by the study coordinator to participants receiving the placebo at the end of visits 2 and 3.
  Memantine: Encapsulated Memantine 10 mg bid (after four-week standard dose titration protocol)
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 73 | 72
ms | -2.52 (96.08) | 0.22 (111.28)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = 2.94, 95% CI 2-sided [-25.32 to 31.20]

8. Secondary Outcome: Safety and Tolerability of the Drug Memantine as Assessed by Change in QTc Interval
Description: Incidence of adverse events was monitored by clinical history, physical examinations, electrocardiograms (ECGs), clinical laboratory tests, the Screen for Childhood Anxiety Related Emotional Disorders (SCARED). Here, we report the analysis of the effect of memantine treatment on QTc intervals because of its clinical importance for this analysis for potential drug toxicity. QTc intervals ≥ 450 ms are generally considered long, and drug-induced QTc interval prolongations ≥ 60 ms are generally considered clinically relevant.
Time Frame: baseline and 16 weeks from start of treatment
Population: The analysis population consisted of all participants who started treatment and had good-quality ECGs before and after the start of memantine treatment, whether or not they completed the entire treatment.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 71 | 65
ms | -1.30 (13.51) | -0.11 (12.38)
Statistical Analysis 1: Comparison: Placebo vs Memantine; QTc interval duration was the independent variable, treatment and time were the categorical factors; Test type: Superiority; p = 0.24, ANOVA; Mean Difference (Net) = -3.04

9. Other Pre Specified Outcome: Intellectual Functioning of the Participants as Assessed by Change in Score on the Matrices Subtest of the Differential Ability Scales-II (DAS-II)
Description: This test provides a measure of non-verbal reasoning ability that requires subjects to visually inspect a matrix of 4 or 9 pictures that has a missing piece. Participants have to infer a rule or pattern in the stimuli and select the appropriate response from a range of 4-6 possibilities. Since age norms are not available for individuals older than 17y11m, the ability score will be used as the dependent variable. This is an intermediate score based on Rasch modeling that corrects for different items set being administered to participants. The minimum value of the DAS-II Rasch Score Scale is 0 and the maximum value is 153; higher scores mean better outcomes. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2).
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 0.75 (9.22) | 2.66 (12.12)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Net) = 1.91, 95% CI 2-sided [-1.57 to 5.39]

10. Other Pre Specified Outcome: Linguistic Functioning of the Participants as Assessed by Change in Score on the Test for Reception of Grammar 2nd Edition (TROG-II)
Description: This is a measure of receptive syntax skills (Bishop, 1983). Participants are asked to point to a picture (out of 4) that corresponds to a phrase or sentence spoken by the examiner. The total number of items correct (rather than blocks passed) will be used as the dependent variable, following the administration manual's ceiling rule. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2). The minimum value of the scores is 0 and the maximum value is 40; with higher scores considered to be a better outcome.
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 0.49 (4.01) | 0.89 (3.39)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.51, Mixed Models Analysis; Mean Difference (Net) = 0.40, 95% CI 2-sided [-0.80 to 1.61]

11. Other Pre Specified Outcome: Linguistic Functioning of the Participants as Assessed by Change in Score on the Peabody Picture Vocabulary Test-IV (PPVT-IV)
Description: This is a measure of receptive semantics, whereby the participant is asked to point to a picture (out of 4) that corresponds to a word spoken by the examiner. As this test has a 0.85 correlation with composite measures of Verbal IQ (i.e. from the Wechsler Intelligence Scale series), it can be used in conjunction with the Matrices subtest to estimate overall intellectual functioning. The total number of items correct was used as the dependent variable, following the administration manual's rules for basals and ceilings. The values for this measure have been recorded as change in score from baseline (T1) to after the treatment (T2). The minimum value for this scale is 0 and the maximum value is 192, higher scores mean a better outcome.
Time Frame: baseline and 16 weeks from start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 76 | 73
score on a scale | 4.46 (12.96) | 5.63 (16.38)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Net) = 1.17, 95% CI 2-sided [-3.6 to 5.94]

12. Other Pre Specified Outcome: Adaptive/Behavioral Functioning of the Participants as Assessed by Change in Score on the Scales of Independent Behavior-Revised (SIB-R)
Description: This is a measure of adaptive functioning that integrates information from 13 different domains (e.g., gross motor, social interaction, eating, toileting, dressing, personal self-care, etc.). It is in a questionnaire format, which a caregiver can complete while the participant is being tested. Standard scores for all indices will be derived from age norms that extend from birth to age 80, as these were used as dependent variables. We report here on the Broad Independence Score recorded as change in score from baseline (T1) to after the treatment (T2). The minimum value of the SIB-R Score Scale in this study was -24 (this number is below 0 because -24 was the minimum value for the worst performing participant in the trial) and the maximum value of this scale is 153; higher scores mean better outcomes.
Time Frame: baseline and 16 weeks from start of treatment
Population: The analysis population consisted of participants who completed 16 weeks of treatment and had neuropsychological assessments at baseline (T1) and after treatment (T2). Note that some participants chose not to undergo the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 67 | 65
score on a scale | 6.88 (16.93) | 3.23 (13.32)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Net) = -3.65, 95% CI 2-sided [-8.91 to 1.61]

ADVERSE EVENTS:
Time Frame: From the beginning to the end of treatment, i.e., 16-18 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov definitions.
Arm/Group | Placebo | Memantine
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/81
Other Adverse Events (participants affected / at risk) | 44/79 | 32/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Memantine (N=81)
Signs and symptoms of upper respiratory viral infection (Infections and infestations) | 12 | 9
Transient dizziness (General disorders) | 6 | 8
Anxiety (Psychiatric disorders) | 4 | 6
Mood changes or irritability (Psychiatric disorders) | 5 | 2
Mood changes or sadness (Psychiatric disorders) | 3 | 3
Oppositional or aggressive behavior (Psychiatric disorders) | 2 | 1
Headache (General disorders) | 3 | 3
Drowsiness (General disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 5
Nausea or vomiting (Gastrointestinal disorders) | 2 | 3
Weakness or fatigue (General disorders) | 1 | 3
Insomnia (General disorders) | 0 | 3
Increase in thyroid-stimulating hormone levels (Endocrine disorders) | 3 | 0 — Clinically significant increase in thyroid-stimulating hormone concentrations in participant with hypothyroidism between screening and follow-up visits
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Increased self-talk (Psychiatric disorders) | 2 | 0
Increased appetite (General disorders) | 2 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Visual hallucinations (Psychiatric disorders) | 0 | 1
Herpes simplex flair-up (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02304302/Prot_SAP_000.pdf